CLINICAL TRIAL: NCT06318806
Title: Towards Remission and Full Recovery From Obsessive-compulsive Disorder: Investigating the Efficacy of Inference-Based Cognitive-Behavioral Therapy When Standard Treatment Has Failed
Brief Title: Towards Remission and Full Recovery From Obsessive-compulsive Disorder
Acronym: RCT2023
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Frederick Aardema,, Full professor, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-3633
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder,; Treatment outcome; Predictors of Outcome; Exposure and Response Prevention; Inference-based Cognitive Behavioral Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: The study is a single site parallel-group randomized-controlled trial with an active run-in treatment. In the first phase of the trial, participants diagnosed with OCD will receive an active run-in treatment consisting of 18 sessions of ERP. In the second phase, non-remitters will be randomly allocated to another 18 sessions of I-CBT or continued treatment with ERP. Non-remission is operationalized in accordance with validated cut-off points established through international consensus and empirical findings (a score of >12 on the YBOCS and a CGI-S rating of 3 or higher (mild to extremely ill) after the run-in treatment with ERP). I-CBT and continued ERP will be followed by a 6-month and 12-month follow-up conforming to current thinking on relapse and recovery in OCD. Treatments will be administered by trained therapists on a weekly one-on-one basis via videoconferencing for the duration of one hour.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure and Response Prevention (Active Comparator): ERP will be delivered in accordance with published guidelines and protocols that employ inhibitory learning principles. Following the creation of a hierarchy of feared situations, patients are encouraged to confront their fears (both during and in-between treatment sessions) while abstaining from engaging in compulsions and other neutralizing strategies (i.e., response prevention). Exercises consist of exposure in vivo (i.e., exposure in real life situations) and/or imaginal exposure that are initially conducted in sessions under the therapist's guidance, and then as daily homework designed by the therapist in collaboration with the patient. In accordance with an inhibitory learning model, rather than focusing on habituation to anxiety, exercises aim to maximize outcomes through expectancy violation, deepened extinction, elimination of safety behaviors during exposure, exposure in multiple contexts, and affect labeling during exposure.
  Interventions: Other: Psychotherapy
- Inference-based Cognitive Behavioral Therapy (Experimental): CBT will be delivered in accordance with published guidelines and protocols that target the dysfunctional reasoning giving rise to obsessional doubts. The first learning point in I-CBT is that the compulsions, anxiety and discomfort are driven by an initial obsessional doubt. The principal focus of treatment is to show that the doubt is 100% irrelevant in the here and now. To this end the reasoning narrative is identified, including the reasoning distortions contained therein, giving undue credibility to the obsessional doubt. The selective nature of the doubt is underlined by showing the client how under most everyday circumstances his/her reasoning is entirely different from the obsessional situation. This stage also educates the client in the thematic nature of the obsessional doubt and how personal themes dictate the idiosyncratic nature of the person's obsession. The final stage of therapy consists of training the client in the proper use of the senses.
  Interventions: Other: Psychotherapy

INTERVENTIONS:
Other: Psychotherapy — Psychotherapy is a type of treatment that can help individuals experiencing mental health conditions and emotional challenges.

SUMMARY:
Obsessive-compulsive disorder (OCD) is a disabling psychiatric illness that is characterized by distressing obsessional thoughts and time-consuming compulsive rituals. Exposure and Response Prevention (ERP) is a first-line psychological treatment of choice that requires patients to face their fears by being exposed to feared stimuli. This treatment has been shown to reduce symptoms in a significant proportion of patients. However, it is considered a difficult treatment and only a minority reach remission. Residual symptoms typically remain, or reappear after treatment, which is a risk for relapse. Inference-based Cognitive Behavioral Therapy (I-CBT) is a promising evidence-based treatment developed to overcome these limitations. I-CBT has already been found to be as effective as ERP and significantly more acceptable and easier to adhere to. There is also evidence that I-CBT is more effective for subgroups of patients. Consequently, the current research project is focused on improving treatments outcomes for those provide those who have previously unable to reach remission of their symptoms with ERP. Following an initial treatment with ERP, those that have been unable to reach remission, will be randomized to either I-CBT or more ERP. It is expected that I-CBT will be significantly more effective than providing patients with more of the same. In addition, the study aims to predict treatment outcome in order to be able to tell in advance which patients do not respond to ERP. The project is designed to maximize beneficial health outcomes with a stepped-care approach to treatment, but also to work towards a more personalized choice by being able to match patients in advance with the treatment that works best for them

DETAILED DESCRIPTION:
Exposure and Response Prevention (ERP) improves symptoms in a significant proportion of patients, but only a minority reach remission after completing ERP (~40%). Also, ERP is a difficult treatment that requires requires deliberate and prolonged exposure to fearful stimuli and is associated with lower levels of acceptability and tolerability. The current trial aims to overcome these limitations with Inference-Based Cognitive-Behavioral therapy (I-CBT) - a specialized form of Cognitive Behavioral Therapy that does not require provoking anxiety through exposure to fearful stimuli. To meet our objective, the current study consists of a randomized controlled trial preceded by a run-in treatment with ERP with a total of 160 patients diagnosed with OCD. Those that fail to reach remission with the run-in treatment (est. 60%) will be randomly allocated to either 18 sessions of ICBT or continued treatment with ERP. Patients will be diagnosed by standardized semi-structured interviews and treatment outcome will be assessed by gold standard clinician rated measurement of severity of symptoms by independent evaluators. For the first hypothesis, it is predicted that I-CBT is superior to continued ERP among those who have previously failed to reach remission with ERP in terms of: (a) greater improvement on our principal continuous outcome measure of OCD severity at post-treatment and follow-up; (b) clinical status at post-treatment and follow-up (treatment response, remission and relapse). For our second hypothesis, it is predicted that I-CBT is more acceptable and tolerable as compared to continued treatment with ERP for those previously unable to benefit sufficiently from ERP. For our third hypothesis, it is predicted that I-CBT is associated with more improvement on our secondary measures of outcome, including a) OC symptom dimensions and negative mood states, b) obsessive beliefs and reasoning processes, and c) psychosocial functioning. For our fourth hypothesis, it is predicted that ERP is associated with a higher frequency of combined treatment refusal and drop-out rates as compared to I-CBT. For our fifth hypothesis, tit is predicted that treatment outcome during ERP and I-CBT is associated with improvements in inferential confusion and feared-self perceptions. The secondary objective of the current proposal is to identify predictors of outcome and to use supervised machine learning to forecast which patients fail to reach remission following initial ERP treatment in order to enable the selection of patients to administer I-CBT as a first-line treatment in the future. Predictors will consist of previously identified risk factors of negative outcome, as well as proposed candidates in the extant literature

ELIGIBILITY:
Inclusion criteria:

1. a primary diagnosis of OCD according to DSM-5 criteria.
2. a score ≥ 18 on the Y-BOCS
3. age ≥ 18.
4. no change in medication during the 8 weeks before treatment for antidepressants (4 weeks for anxiolytics).
5. willingness to keep medication stable while participating in the study.
6. not undergoing a concurrent psychological treatment.
7. access to a computer or phone with internet access.

   Exclusion criteria:
8. evidence of a high level of suicidal ideation, suicidal intent or previous suicide attempts.
9. past or present psychotic or bipolar disorder.
10. neurocognitive disorder, pervasive developmental disorder or intellectual disability of a severity judged to significantly interfere with treatment and/or requiring treatment first.
11. substance abuse disorder of a severity judged to significantly interfere with treatment and/or requiring treatment first.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale -2 (Y-BOCS-2) | Baseline, change after 9 weeks of treatment, 18 weeks of treatment, change in phase 2 after 9 weeks of treatment, change in phase 2 after 18 weeks of treatment, change after 6-month follow-up, change after 12-month follow-up
  he Yale-Brown Obsessive-Compulsive Scale - 2 is the instrument of choice to assess obsessive compulsive symptoms and severity. Total scores on the measure range from 0 to 40 with higher scores indicating more severe symptoms.
Clinical Global Impression Scale (CGI) | Baseline, change after 9 weeks of treatment, 18 weeks of treatment, change in phase 2 after 9 weeks of treatment, change in phase 2 after 18 weeks of treatment, change after 6-month follow-up, change after 12-month follow-up
  The clinical global impression rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. Scores on the measure range from 1 to 7 with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Vancouver Obsessional Compulsive Inventory (VOCI) | Baseline, change after 9 weeks of treatment, 18 weeks of treatment, change in phase 2 after 9 weeks of treatment, change in phase 2 after 18 weeks of treatment, change after 6-month follow-up, change after 12-month follow-up
  The Vancouver Obsessional Compulsive Inventory (VOCI) to assess a broad spectrum of OCD symptoms and associated personality characteristics.It is a 55-item self-report measure to assess a broad spectrum of OCD symptoms. Total scores on the measure range from 0 to 220 with higher scores indicating more severe symptoms.
Beck Depression Inventory (BDI) | Baseline, change after 9 weeks of treatment, 18 weeks of treatment, change in phase 2 after 9 weeks of treatment, change in phase 2 after 18 weeks of treatment, change after 6-month follow-up, change after 12-month follow-up
  The Beck Depression Inventory (BDI) is a standard 21-item measure to assess depressive symptoms.. Total scores on the measure range from 0 to 63 with higher scores indicating more severe symptoms.
Beck Anxiety Inventory (BAI) | Baseline, change after 9 weeks of treatment, 18 weeks of treatment, change in phase 2 after 9 weeks of treatment, change in phase 2 after 18 weeks of treatment, change after 6-month follow-up, change after 12-month follow-up
  The Beck Anxiety Inventory (BAI) is a standard 21-item anxiety symptom checklist rating anxiety symptom intensity for the last week on a 0-3 scale. Total scores on the measure range from 0 to 63 with higher scores indicating more severe symptoms.
Inferential Confusion Questionnaire (ICQ) | After baseline before treatment, change after 9 weeks of treatment, 18 weeks of treatment, change in phase 2 after 9 weeks of treatment, change in phase 2 after 18 weeks of treatmen
  The ICQ is a 30-item questionnaire measuring dysfunctional reasoning processes. Total scores on the measure range from 0 to 180 with higher scores indicating higher levels of dysfunctional reasoning.
Dysfunctional Reasoning Processes Task (DRPT) | After baseline before treatment, change after 18 weeks of treatment, change in phase 2 after 18 weeks of treatment
  The Dysfunctional Reasoning Processes Task (DRPT) is a task based measure of inferential confusion. Total scores on the measure range from 0 to 21 with higher scores indicating higher levels of dysfunctional reasoning.
Fear of Self Questionnaire-Multidimensional Version | After baseline before treatment, change after 18 weeks of treatment, change in phase 2 after 18 weeks of treatment
  The Fear of Self Questionnaire (FSQ-MV) is a measure of feared self-perceptions. Total scores on the measure range from 0 to 180 with higher scores indicating higher levels of fear of self.
Obsessive Beliefs Questionnaire (OBQ-20) | After baseline before treatment, change after 18 weeks of treatment, change in phase 2 after 18 weeks of treatment
  The Obsessive Beliefs Questionnaire (OBQ-20) is a 20-item measure developed by the Obsessive Compulsive Cognitions Working Group measuring obsessive compulsive beliefs(over-responsibility/over-estimation of threat, intolerance of uncertainty/over-importance of thought, control of thoughts/perfectionism). Total scores on the measure range from 0 to 140 with higher scores indicating more higher endorsement of obsessive beliefs.
Brunnsviken Brief Quality of Life Scale (BBQ) | After baseline before treatment, change after 18 weeks of treatment, change in phase 2 after 18 weeks of treatment
  The Brunnsviken Brief Quality of Life Scale (BBQ) is a 12 item self-report questionnaire that assesses subjective quality of life across six life areas: Leisure, View on Life, Creativity, Learning, Friends and Friendship, and View on Self. Total scores on the measure range from 0 to 48 with higher scores indicating a better quality of life.
Sheehan Disability Scale | Baseline, change after 9 weeks of treatment, 18 weeks of treatment, change in phase 2 after 9 weeks of treatment, change in phase 2 after 18 weeks of treatment, change after 6-month follow-up, change after 12-month follow-up
  The Sheehan Disability Scale measures the functional capacity at the professional, social and family level of the participant/patient. Total scores on the measure range from 0 to 30 with higher scores indicating more functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Aardema, PhD, Principal Investigator — Institut universitaire en santé mentale de Montréal
Locations (1):
- Institut universitaire en santé mentale de Montréal, Montreal, Quebec, Canada